CLINICAL TRIAL: NCT03320707
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-54767414 (Daratumumab) in Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-54767414 (Daratumumab) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108356; 54767414EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-10-11; First posted 2017-10-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daratumumab (Experimental): Participants will receive a single subcutaneous (SC) dose of daratumumab in each of first 7 dose cohorts. Doses will be escalated based on review of pharmacokinetic, pharmacodynamic, and safety data of previous cohort. Participants in Cohort 8 will receive single SC daratumumab formulation containing recombinant human hyaluronidase (rHuPH20).
  Interventions: Drug: Daratumumab; Drug: rHuPH20
- Placebo (Placebo Comparator): Participants will receive placebo as a single SC dose in each of first 7 cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daratumumab — Single SC dose of daratumumab will be administered in each of 8 dose cohorts.
  Other Names: JNJ-54767414
  Arms: Daratumumab
Drug: Placebo — Placebo liquid will be administered as SC dose in each of first 7 dose cohorts.
  Arms: Placebo
Drug: rHuPH20 — Participants in Cohort 8 will receive single SC dose of rHuPH20 as a part of daratumumab formulation.
  Arms: Daratumumab

SUMMARY:
The purpose of this study is to assess the safety and tolerability of daratumumab following a single subcutaneous (SC) administration in healthy participants and to determine whether premedication with corticosteroids is required to improve the tolerability of SC administration of daratumumab in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body weight in the range of 50 to 100 kilogram (kg), inclusive, and have a body mass index (BMI) of 19 to 30 kilogram per meter square (kg/m^2), inclusive, at screening and Day -1
* Must be otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and Day -1
* Must be otherwise healthy on the basis of clinical laboratory tests performed at screening and Day -1
* A woman must not be of childbearing potential
* Must be a non-smoker or tobacco user or 3 months prior to screening

Exclusion Criteria:

* Pregnant or breastfeeding while enrolled in this study or within 20 weeks after the dose of study treatment
* History of or currently has any clinically significant medical illness or medical disorders the investigator considers significant, including, but not limited to immune deficiency state, liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has a history of malignancy before screening. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk of recurrence
* Active acute or chronic infection (including chronic recurrent or invasive candidiasis) or diagnosed latent infection
* Has had a Bacille Calmette-Guérin (BCG) vaccination within 12 months of screening and/or plan to receive a BCG vaccine within 12 months after the administration of study treatment
* Has experienced a recent single dermatomal herpes zoster eruption within the past 6 months
* Has a history of multi-dermatomal herpes zoster or central nervous system (CNS) zoster within the past 5 years
* Has received prescription medications within 14 days prior to study treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Treatment-Emergent Adverse Event (TEAEs) by Severity Through Day 141 Versus Placebo | Up to Day 141
  The safety and tolerability of daratumumab following a single subcutaneous (SC) administration in healthy participants will be assessed.
Proportion of Participants With TEAEs by Serious Adverse Events (SAEs) Through Day 141 Versus Placebo | Up to Day 141
  The safety and tolerability of daratumumab following a single subcutaneous (SC) administration in healthy participants will be assessed.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 predose through Day 141
  Cmax is the maximum observed plasma concentration.
Time to the Maximum Observed Plasma Concentration (Tmax) | Day 1 predose through Day 141
  Tmax is defined as actual sampling time to reach maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to the Time Corresponding to the Last Quantifiable Serum Concentration (AUC [0-last]) | Day 1 predose through Day 141
  AUC (0-last) is the area under the plasma concentration-time curve from time zero to the time corresponding to the last quantifiable serum concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinity With Extrapolation of the Terminal Phase (AUC[0- infinity]) | Day 1 predose through Day 141
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinity with extrapolation of the terminal phase, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Number of Participants With Anti-daratumumab Antibodies | Day 1 predose through Day 141
  Number of participants who test positive for anti-daratumumab antibodies will be reported.
Number of Participants With Anti-recombinant Human Hyaluronidase (rHuPH20) Antibodies | Day 1 predose through Day 141
  Number of participants who test positive for anti-rHuPH20 antibodies will be reported.
Percentage of CD38 Expression Levels and CD38 Expressing Cell Counts Measured by Flow Cytometry | Day 1 predose through Day 141
  The cluster of differentiation (CD) 38 expression levels and CD38 expressing cell counts, as measured by flow cytometry, will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States